CLINICAL TRIAL: NCT05784337
Title: Evaluation of the Efficacy and Safety of the Mi-thos® Transcatheter Mitral Valve Replacement System in Patients With Severe Mitral Valve Disease at High Surgical Risk(First-in-Man Study)
Brief Title: Mi-thos® Transcatheter Mitral Valve Replacement(First-in-Man Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai NewMed Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mi-thos-FIM
Record Dates: First submitted 2023-03-12; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mi-thos® Transcatheter Mitral Valve Replacement System (Experimental): Transcatheter mitral valve replacement with the Mi-thos® valve and transcatheter delivery system
  Interventions: Device: Mi-thos® Transcatheter Mitral Valve Replacement System

INTERVENTIONS:
Device: Mi-thos® Transcatheter Mitral Valve Replacement System — Transcatheter Mitral Valve Replacement

SUMMARY:
To evaluate the effectiveness and safety of the Mi-thos® Transcatheter Mitral Valve Replacement System in the treatment of patients with moderate or greater mitral regurgitation who are at high risk for conventional surgery, or who are not candidates for conventional surgery.

DETAILED DESCRIPTION:
The Mi-thos® study is a single-arm, prospective, safety and performance clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Severe mitral regurgitation ≥ 3+;
* Patients with an STS score >8 or who have been evaluated by a cardiothoracic surgeon as high risk for conventional surgery or who cannot tolerate conventional open-heart surgery;
* Age ≥ 65 years old;
* Life expectancy > 12 months;
* Patients sign an informed consent form.

Exclusion Criteria:

* Previous cardiac mitral valve surgery;
* Active infections requiring antibiotic therapy;
* Clinically significant untreated Coronary Artery Disease (CAD);
* Pulmonary hypertension （Pulmonary systolic pressure > 70 mmHg）;
* Patients with severe right heart failure;
* Left ventricular ejection fraction <25%;
* Diagnosis of hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis;
* Dialysis patient;
* Patients with severe coagulopathy;
* Patients with contraindications to anticoagulant drugs;
* Patients with stroke or transient ischemic within 30 days;
* Echocardiography found any intracardiac mass, left ventricle or atrial thrombus;
* Patients who require surgery or interventional therapy for other valvular lesions;
* Patients with severe macrovascular disease requiring surgical treatment;
* Patients with more than 70% of carotid stenosis;
* To be allergic to contrast agents, nickel-titanium memory alloys or bovine-derived products;
* Patients with severe neurological disorders affecting cognitive ability;
* Life expectancy < 12 months;
* Patients with severe thoracic deformities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Technical success | immediate post-surgical
  All of the following must be present:
  I. Absence of procedural mortality; and II. Successful access, delivery, and retrieval of the device delivery system; and III. Successful deployment and correct positioning of the first intended device; and IV. Freedom from emergency surgery or reintervention related to the device or access procedure

SECONDARY OUTCOMES:
Rate of all-cause mortality | 30 days
  All-cause mortality after TMVR
Rate of Severe adverse event | 30 days
  Severe adverse events rate after TMVR
Device success | 30 days
  All of the following must be present:
  I. Absence of procedural mortality or stroke; and II. Proper placement and positioning of the device; and III. Freedom from unplanned surgical or interventional procedures related to the device or access procedure; and
  IV. Continued intended safety and performance of the device, including:
  A. No evidence of structural or functional failure B. No specific device-related technical failure issues and complications C. Significant alterations in mitral valve hemodynamics (MR≤moderate/EOA≥ 1.5 cm2/mean transmitral gradient < 5 mmHg/no paravalvular MR associated hemolysis)
Procedural success | 30 days
  All of the following must be present:
  I. Device success, and
  II. Absence of major device or procedure related serious adverse events, including:
  A. Death B. Stroke C. Life-threatening bleeding (MVARC scale) D. Major vascular complications E. Major cardiac structural complications F. Stage 2 or 3 acute kidney injury (includes new dialysis) G. Myocardial infarction or coronary ischaemia requiring PCI or CABG H. Severe hypotension, heart failure, or respiratory failure requiring intravenous pressors or invasive or mechanical heart failure treatments I. Any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention
Incidence of arrhythmia or conduction block | 30 days
  Incidence of arrhythmia or conduction block after TMVR

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Air Force Medical University, Xi’an, Shanxi